CLINICAL TRIAL: NCT00842413
Title: What Part Does the Premotor Cortex Play in Subjective Visual Perception and in the Perception of Others' Actions?
Brief Title: Investigating the Role of the Premotor Cortex in Higher Cognitive Functions
Status: Terminated | Type: Observational
Why Stopped: not enough enrollment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick Vacher, Clinical Research Department of Developpement
Other Study IDs: P060605
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2008-11

CONDITIONS: Brain Injury; Chronic
Keywords: Prefrontal cortex; visual consciousness; focal lesions; action perception
MeSH Terms: conditions — Brain Injuries; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: The study compares brain-damaged patients with healthy ones on two psychophysical tasks.
- 2: The study does not intervene on the brain-damaged patients, it merely compares their behaviour with that of healthy patients on a range of psychophysical tasks.

SUMMARY:
This project aims at understanding better the role of the frontal lobe of the brain in our capacity to perceive visual information consciously, and also, in our capacity to perceive others' actions. It includes a test where we ask subjects to detect visual information in front of a computer screen, and another test where we ask them to imitate finger movements.

DETAILED DESCRIPTION:
This project is a twofold exploration of the functions of the premotor cortex, concerning, on the one hand, its role in conscious visual perception, and on the other hand, the part it may play in the perception and imitation of other people's movements. Healthy subjects will be compared with subjects suffering from focal lesions within the premotor cortex, on two tasks: in the first task, the subjects will have to make a decision concerning the absence or presence of a visual item in their field of vision. They will make (virtual) bets based on the subjective certainty of their perceptions - they will be told that these bets are purely virtual, and will not result in any financial gain or loss. This study will help us understand the contribution of the prefrontal cortex to subjective weighing of perceptual certainty. In the second task, the subjects will imitate a finger movement, based either on a fixed picture, or on a short motion picture. Previous studies have shown that whether the movement is copied from a fixed picture or a moving picture changes reaction times and types of mistakes. Neuroimaging studies have shown that a premotor area is involved in this effect. The comparison of brain-damaged and healthy subjects will tell us what exactly the contribution of the prefrontal consists in.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects chosen from a pool of adult subjects, recruited through ads.
* In the second group, the subjects are recruited from a pool of brain-damaged patients treated at the hospital de la Pitié-Salpétrière. They must suffer from a focal lesion in the prefrontal cortex.

Exclusion Criteria:

* For the healthy group: any previous brain-related medical history.
* Widespread brain-damage, extending beyond the prefrontal cortex, that is to say, lesions that are not really focal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The visual pereption of subjects willl be studied, but no attempt will be made at modifying it, or treating any problem that they might have.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2007-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Levy, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital de la Pitié-Salpétrière, Paris, France